CLINICAL TRIAL: NCT05180799
Title: A Phase 1/2 Study of BA3071 in Patients With Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: BioAtla, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BA3071-001
Record Dates: First submitted 2021-12-14; First posted 2022-01-06 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2024-10

CONDITIONS: NSCLC; Melanoma
Keywords: metastatic; cancer; First Line Melanoma; First Line NSCLC; 1L NSCLC; Treatment Refractory Melanomas; Nonsquamous Stage IV; Nonsquamous recurrent; 1L NSCLC; Systemic Treatment Naive; Nonsquamous Stage IIB; Nonsquamous Stage IIIA; KRAS; STK11; KEAP1; PD-L1 tumor proportion score (TPS) <1%
MeSH Terms: conditions — Melanoma; Neoplasm Metastasis; Neoplasms | interventions — Nivolumab; pembrolizumab; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- BA3071 (Experimental): Conditionally active biologic (CAB) antibody that binds to CTLA-4
  Interventions: Biological: BA3071
- Combination Therapy (Experimental): Conditionally active biologic (CAB) antibody that binds to CTLA-4 with PD-1 inhibitor
  Interventions: Biological: BA3071; Biological: Nivolumab; Biological: Pembrolizumab
- Combination Therapy + Chemotherapy (Experimental): Conditionally active biologic (CAB) antibody that binds to CTLA-4 with PD-1 inhibitor + Chemotherapy
  Interventions: Biological: BA3071; Biological: Pembrolizumab; Drug: Pemetrexed (Alimta)
- Neoadjuvant Combination Therapy + Chemotherapy (Experimental): Conditionally active biologic (CAB) antibody that binds to CTLA-4 with PD-1 inhibitor + Chemotherapy prior to surgical resection
  Interventions: Biological: BA3071; Biological: Pembrolizumab; Drug: Pemetrexed (Alimta)

INTERVENTIONS:
Biological: BA3071 — Conditionally active biologic (CAB) antibody that binds to CTLA-4
Biological: Nivolumab — Humanized, immunoglobulin G4 (IgG4)-variant mAb against PD-1
  Arms: Combination Therapy
Biological: Pembrolizumab — Humanized antibody, immunoglobulin G4, with a variable region against the human PD-1 receptor
  Arms: Combination Therapy; Combination Therapy + Chemotherapy; Neoadjuvant Combination Therapy + Chemotherapy
Drug: Pemetrexed (Alimta) — pemetrexed with either cisplatin or carboplatin
  Arms: Combination Therapy + Chemotherapy; Neoadjuvant Combination Therapy + Chemotherapy

SUMMARY:
The objective of this study is to assess safety and efficacy of BA3071 in solid tumors

DETAILED DESCRIPTION:
This is a multi-center, open-label study designed to evaluate the safety, tolerability, PK, immunogenicity, and antitumor activity of BA3071. Phase 2 is open and currently recruiting patients with:

1. Melanoma - 1L
2. nonsquamous or recurrent NSCLC (Type IIB, IIIA, IV) with single or any combination of the following mutations: KRAS mutation STK11 mutation KEAP1 mutation PD-L1 tumor proportion score (TPS) <1%

ELIGIBILITY:
Inclusion Criteria:

* Patients must have measurable disease.
* Age ≥ 18 years
* CLTA-4 blocking-antibody naïve
* Adequate renal function
* Adequate liver function
* Adequate hematological function
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Patients must have single or any combination of the following mutations: KRAS, STK11, KEAP1 and/or PD-L1 TPS <1%
* Patients must be eligible for surgery (NSCLC Stage IIB-IIIA only)

Exclusion Criteria:

* Patients must not have clinically significant cardiac disease.
* Patients must not have known non-controlled CNS metastasis.
* Patients must not have a history of ≥ Grade 3 allergic reactions to mAb therapy as well as known or suspected allergy or intolerance to any agent given during this study.
* Patients must not have had major surgery within 4 weeks before first BA3071 administration.
* Patients must not have known human immunodeficiency virus (HIV) infection, active hepatitis B and/or hepatitis C.
* Patients must not be women who are pregnant or breast feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2022-08-03 (Actual); Primary Completion 2025-03-19 (Actual); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Assess dose limiting toxicity as defined in the protocol | Up to 24 months
  Phase 1: Safety Profile
Assess maximum tolerated dose as defined in the protocol | Up to 24 months
  Phase 1: Safety Profile
Frequency and severity of AEs and/or SAEs | Up to 24 months
  Phase 1 and 2: Safety Profile
Confirmed overall response rate (ORR) per RECIST v1.1 | Up to 24 months
  Phase 2: Efficacy

SECONDARY OUTCOMES:
Phase 1: Pharmacokinetics | Up to 24 months
  Plasma concentrations of ADC
Phase 1: Pharmacokinetics | Up to 24 months
  Plasma concentrations of total antibody
Phase 1: Pharmacokinetics | Up to 24 months
  Plasma concentrations of MMAE
Peak Plasma Concentration (Cmax) | Up to 24 months
  Phase 1: Pharmacokinetics
Area under the plasma concentration versus time curve (AUC) | Up to 24 months
  Phase 1: Pharmacokinetics
Confirmed best overall response (BOR) | Up to 24 months
  Phase 1 and 2: Efficacy
Confirmed overall response rate (ORR) | Up to 24 months
  Phase 2: Efficacy
Disease control rate (DCR) | Up to 24 months
  Phase 1 and 2: Efficacy
Time to response (TTR) | Up to 24 months
  Phase 1 and 2: Efficacy
Overall survival (OS) | Up to 24 months
  Phase 1 and 2: Efficacy
Percent change from baseline in target lesion sum of diameters. | Up to 24 months
  Phase 1 and 2: Efficacy
Duration of response (DOR) | Up to 24 months
  Phase 1 and 2: Efficacy
Progression-free survival (PFS) | Up to 24 months
  Phase 1 and 2: Efficacy

CONTACTS AND LOCATIONS:
Locations (12):
- United States (9):
  - The Angeles Clinic and Research Institute, Los Angeles, California
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - Piedmont West, Atlanta, Georgia
  - Northwest Cancer Centers, Dyer, Indiana
  - Morristown Medical Center/Atlantic Health System, Morristown, New Jersey
  - Icahn School of Medicine at Mt. Sinai, New York, New York
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Providence Cancer Institute, Portland, Oregon
  - University of Utah Huntsman Cancer Institute, Salt Lake City, Utah
- Australia (3):
  - Border Medical Oncology Research Unit at Albury Wodonga Regional Cancer Centre, Albury, New South Wales
  - Cancer Care Foundation, Miranda, New South Wales
  - Cancer Research South Australia, Adelaide, South Australia

IPD SHARING:
Plan to Share IPD: Undecided